CLINICAL TRIAL: NCT01947075
Title: Etiologies of Acute Febrile Illness Among Adults Attending an Outpatient Department in Dar es Salaam
Brief Title: Etiologies of Fever Among Adults in Dar es Salaam
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Principal Investigator, Valérie D'Acremont, Investigator, Swiss Tropical & Public Health Institute
Other Study IDs: Fever Study; Adult Fever Study (Other: SwissTPH)
Record Dates: First submitted 2013-09-13; First posted 2013-09-20 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Acute Febrile Illnesses
Keywords: Fever; Tanzania; Pneumonia; HIV; Diabetes; Indoor Air Pollution
MeSH Terms: conditions — Fever; Pneumonia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Whole blood Serum Sputa Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adults with fever: Every adult with fever will be screened for different infectious diseases and for nasopharyngeal respiratory viruses and bacteria
- Healthy volonteers: For every adult with fever included with a diagnosis of pneumonia, a healthy volunteer will be included. These healthy volunteers will be screened for nasopharyngeal respiratory viruses and bacteria.

SUMMARY:
Following the decline of malaria in Sub-Saharan Africa, clinicians face febrile patients in whom an alternative diagnosis has to be made. This situation has led to an overuse of antibiotics by clinicians. It is crucial to increase knowledge on etiologies and risk factors of outpatient febrile illness in order to improve their management.

This present proposal aims to investigate the etiologies of fever among adult patients attending an outpatient department in urban Tanzania. It also aims to assess the clinical significance of nasopharyngeal (NP) respiratory viruses and bacteria documentation in this setting. Third, it aims to compare the spectrum of infections in this population with that of children included in the same setting in a previous study. The last objective is to assess diabetes mellitus (DM) as a risk factor for infection and exposure to indoor air pollution (IAP) as a risk factor for acute respiratory infections (ARI) in adults in Tanzania.

The investigators hypothesize that acute respiratory infections are the main cause of adult febrile illness in a urban low-income setting and that use of quantitative molecular assays on naso-oropharyngeal samples can improve the diagnosis of pneumonia. The investigators also think that the spectrum of infections is different between children and adults, mainly due to a high HIV prevalence in adults. The investigators also hypothesize that experiencing IAP and/ or DM is a risk factor for infections in adults.

ELIGIBILITY:
Inclusion Criteria:

* Temperature >=38°C
* History of fever for less than 8 days
* First consultation for the present problem

Exclusion Criteria:

* Refusal of HIV screening
* Main complaint is injury or trauma
* Antibiotic treatment in the last 7 days
* Within 6 weeks after delivery
* Hospitalization during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every consecutive adult with temperature ≥38°C attending the outpatient department of Mwananyamala Hospital will be screened for inclusion. Additional inclusion criteria are fever of ≤1 week duration and first consultation for the present problem. Exclusion criteria are refusal of HIV screening, main complaint is injury or trauma, antibiotic treatment during the previous week (apart from cotrimoxazole prophylaxis), delivery within the previous 6 weeks and hospitalization during the last month. Medical history will be taken (including exposure to IAP) and clinical examination will be done in a standardized way.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with each disease among all febrile patients, overall and stratified by HIV status | 1 year
  Description of the distribution of causes of fever based on pre-defined case definitions for each disease.

SECONDARY OUTCOMES:
Proportion of febrile patients with acute respiratory infection infected with a certain respiratory pathogen, compared to the proportion of healthy controls infected with the same pathogen. | 1 year
  Nasopharyngeal respiratory viruses and bacteria documentation (presence/absence as well as pathogen loads) will be compared between patients with acute respiratory infection and a control group of healthy volunteers

OTHER OUTCOMES:
Strength of association between each febrile disease and diabetes mellitus and between acute respiratory infections and indoor air pollution | 1 year
  Screening of diabetes mellitus and screening of exposure to indoor air pollution will be performed among patients with fever. The strength of association between diabetes and each type of febrile disease and exposure to indoor air pollution and acute respiratory infections will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie D'Acremont, MD PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Mwananyamala Hospital, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Boillat-Blanco N, Klaassen B, Mbarack Z, Samaka J, Mlaganile T, Masimba J, Franco Narvaez L, Mamin A, Genton B, Kaiser L, D'Acremont V. Dengue fever in Dar es Salaam, Tanzania: clinical features and outcome in populations of black and non-black racial category. BMC Infect Dis. 2018 Dec 12;18(1):644. doi: 10.1186/s12879-018-3549-z. PMID 30541456
- [Derived] Boillat-Blanco N, Mbarack Z, Samaka J, Mlaganile T, Mamin A, Genton B, Kaiser L, Calandra T, D'Acremont V. Prognostic value of quickSOFA as a predictor of 28-day mortality among febrile adult patients presenting to emergency departments in Dar es Salaam, Tanzania. PLoS One. 2018 Jun 14;13(6):e0197982. doi: 10.1371/journal.pone.0197982. eCollection 2018. PMID 29902174